CLINICAL TRIAL: NCT04431011
Title: Layer-specific Contribution to Consolidation of Skill Learning in the Primary Motor Cortex
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200105; 20-N-0105
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10-27

CONDITIONS: Normal Physiology
Keywords: Healthy; Learning Consolidation; Brain; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Healthy right-handed participants aged 18-50

SUMMARY:
Background:

Training in a new motor skill often involves periods of active practice and periods of rest. During early motor skill learning, improvements in performance usually happen during the short rest periods between practice sessions. Researchers want to use improved imaging techniques to study the contributions of specific parts of the brain to how people learn and retain movement skills.

Objective:

To learn the part played by different layers in the brain in retaining a newly learned movement skill.

Eligibility:

Healthy, right-handed, English-speaking people age 18-50.

Design:

Participants will be screened with:

* Medical and neurological history
* Medicine review
* Physical exam
* Neurological exam.

Participants may have 2 magnetic resonance imaging (MRI) scans of the brain. During the MRI, they will lie in the scanner. The scanner makes noise. They will get earplugs.

Participants will have behavior testing. A specific order of keys will be displayed on a computer screen. Participants will practice typing the keys with their left hand 36 times (in 10-second blocks). They will repeat this test with a random order of keys.

Participants will see single numbers displayed one after the other on the computer screen. They will make single tap responses using the finger that corresponds with the number on the screen.

Participants will have up to 4 study sessions. Each session will take about 5 hours.

DETAILED DESCRIPTION:
Study Description:

Training on a novel motor skill often involves periods of active practice interspersed with periods of rest. During early motor skill learning, performance improvements develop primarily during short offline rest periods that occur between practice blocks. These performance gains during rest have been referred to as 'micro-offline consolidation'. Primary motor cortex (M1) is a crucial contributor to skill consolidation, however, due to the poor spatial specificity and vascular biases of available imaging methods, the specific neural mechanisms of consolidation in M1 are not known. Recent innovations in functional magnetic resonance imaging (fMRI) have made it possible to measure functional changes across cortical layers. This study will use these techniques to investigate the contributions of specific cortical layers in M1 to motor skill learning and consolidation.

Objectives:

The primary aim is to determine the correlation between activity in superficial M1 cortical layers and behavioral gains during microoffline rest periods. Additionally, we will evaluate the role of superficial and deep cortical layers of M1 in the consolidation of motor skill learning. To address this question, we will measure neural activations across cortical laminae in M1 while participants consolidate a newly acquired motor skill.

Endpoints:

The primary endpoint measures will be: 1) activity in superficial M1 cortical layers during micro-offline rest periods, which will be measured using vascular space occupancy (VASO) MR imaging and 2) behavioral gains during micro-offline rest periods measured as correct sequence typing speed (sequences per second). The secondary endpoint measure will be the ratio of activity between superficial and deep M1 layers during practice and during rest periods compared to pre-learning and to post-learning rest and the localizing random sequence.

Exploratory endpoints will include other fMRI measures that may relate learning with layer activity. For example, we will use multivoxel pattern analysis (MVPA) of activation data to: (a) gain insight into the presence of layer-specific reactivation of sequence task performance during rest periods; and (b) investigate whether this reactivation predicts learning.

Study Population:

45 Healthy participants (18-50 years of age)

Phase:

N/A

Description of Sites/Facilities Enrolling Participants:

This protocol utilizes the NIH Clinical Center Outpatient Clinic, and NMRF core facilities.

Intervention Study Duration:

24 months

Participant Duration:

Approximately 2-5 hours per session, for up to 4 sessions over a 1-4-day time period.

Study Description:

Training on a novel motor skill often involves periods of active practice interspersed with periods of rest. During early motor skill learning, performance improvements develop primarily during short offline rest periods that occur between practice blocks. These performance gains during rest have been referred to as "micro-offline consolidation". Primary motor cortex (M1) is a crucial contributor to skill consolidation; however, due to the poor spatial specificity and vascular biases of available imaging methods, the specific neural mechanisms of consolidation in M1 are not known. Recent innovations in functional magnetic resonance imaging (fMRI) have made it possible to measure functional changes across cortical layers. This study will use these techniques to investigate the contributions of specific cortical layers in M1 to motor skill learning and consolidation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-50
* English speaking
* Right-hand dominance (>74 on Edinburgh Handedness Inventory)
* Normal neurological examination
* Willing and able to provide informed consent

EXCLUSION CRITERIA:

* HCPS-affiliated NIH staff (i.e. - staff from our section).
* Current pregnancy
* Current or past history of use of antiepileptic drugs
* Contraindications for MRI (such as certain implants, metal fragments or devices in the body) as determined by the screening clinician
* Severe or progressive neurological, psychological or medical condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy right-handed adults aged 18-50
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
The primary aim is to determine the role of superficial and deep cortical layers of M1 in the consolidation of motor skill learning. | 4 years
  To address this question, we will measure neural activations across cortical laminae in M1 while participants consolidate a newly acquired motor skill.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-N-0105.html